CLINICAL TRIAL: NCT04771104
Title: The Effect of Induced Hyperammonaemia on Sleep and Melanopsin-mediated Pupillary Light Response in Patients With Liver Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Peter Nissen Bjerring, Consultant hepatologist, associate professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H15000210
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Hepatic Encephalopathy; Liver Cirrhosis; Sleep Disturbance
MeSH Terms: conditions — Hepatic Encephalopathy; Liver Cirrhosis; Parasomnias

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allocated to intervention at first experimental day (Active Comparator)
  Interventions: Dietary Supplement: Amino Acid Challenge (AAC)
- Allocated to intervention at second experimental day (Placebo Comparator)
  Interventions: Dietary Supplement: Amino Acid Challenge (AAC)

INTERVENTIONS:
Dietary Supplement: Amino Acid Challenge (AAC) — The AAC contains 54 g banana flavoured amino acid mixture added 200-300 mL of water. The AAC simulates the composition of haemoglobin in approximately 400 mL of blood.

SUMMARY:
Sleep disturbances are common among patients with liver cirrhosis, but the reasons are not well understood. In this project the investigators evaluated whether an increase in blood ammonia in patients with cirrhosis had an impact on sleep quality and the function of retinal ganglion cells measured by pupillary response to blue light.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of Child Pugh Class A or B cirrhosis
* Written informed consent
* >20 and <80 years of age

Exclusion Criteria:

* Misuse of alcohol in the preceding 6 months,
* Episodes of hepatic decompensation leading to in-patient admissions during the previous month
* History or clinical signs of overt HE or severe sleep-wake disturbances
* On anti-HE treatment (lactulose, rifaximin, Hepa-Merz, Generaid, Bramino)
* History of significant head injury
* Neurological/psychiatric comorbidity needing medical treatment
* Taking neuroactive medication/medication known to affect sleep
* Travel across more than two time zones in the preceding 3 months
* Shift work in the preceding 5 years
* Contraindications for arterial puncture (negative collateral circulation test, wrist infection or vascular abnormalities).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-09 (Actual); Study Completion 2018-01-22 (Actual)

PRIMARY OUTCOMES:
Difference in the late post-illumination pupillary response after intervention compared to placebo | 12 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of gastroenterology and hepatology, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kann AE, Ba-Ali S, Seidelin JB, Larsen FS, Hamann S, Bjerring PN. The effect of induced hyperammonaemia on sleep and melanopsin-mediated pupillary light response in patients with liver cirrhosis: A single-blinded randomized crossover trial. PLoS One. 2022 Sep 28;17(9):e0275067. doi: 10.1371/journal.pone.0275067. eCollection 2022. PMID 36170326